CLINICAL TRIAL: NCT01249235
Title: Prospective Randomized Controlled Trial Comparing Bandage Contact Lens and Oral Analgesics Versus Patching and Oral Analgesics for Pain Following Pterygium Surgery
Brief Title: Bandage Contact Lens and Oral Analgesics Versus Patching and Oral Analgesics for Pain Following Pterygium Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Allan Slomovic, Toronto Western Hospital, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB-10-0538
Record Dates: First submitted 2010-11-22; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-10

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Transdermal Patch

ARMS (2):
- Patch (Active Comparator): The operative eye will be patched.
  Interventions: Procedure: Patch or bandage contact lens
- Bandage Contact Lens (Experimental): The operative eye will have a bandage contact lens
  Interventions: Procedure: Patch or bandage contact lens

INTERVENTIONS:
Procedure: Patch or bandage contact lens — Patients will be given a patch or a bandage contact lens at the conclusion of pterygium excision surgery.

SUMMARY:
The purpose of this study is to determine if patching the eye or a bandage contact lens along with Tylenol #3 is more effective for pain control following pterygium surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary pterygium (no previous surgeries or radiotherapy) requiring excision due to ocular discomfort or disruption in vision
* Size of pterygium greater than 2.5 mm over the cornea (pterygia smaller than this do not result in much postoperative eye pain)
* Ability to understand the nature of the procedure and to complete all measurement requirements
* Adults (age greater than 18)

Exclusion Criteria:

* Ocular surface disease apart from pterygium (such as severe dry eye, corneal disease, scarring from previous infection, radiotherapy, inflammatory diseases or trauma)
* Patients who have had previous ocular surface surgery
* Contraindications to local anesthetics (such as known allergy)
* Pregnancy (as the risk to the fetus with the use of topical antibiotic drops and local anesthetics are not known)
* Patients already on systemic analgesics for any other reason (such as rheumatoid arthritis)
* Allergy to codeine (in order to standardize the systemic analgesic used so that we can compare the effect of bandage contact lens versus 24 hour patching)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Score | 1 week

SECONDARY OUTCOMES:
Sensitivity to light, tearing, foreign body sensation | 1 week
Postoperative Complications | 1 week
  Difficulty removing the bandage lens, the bandage lens has fallen out, graft dislocation
Number of Tylenol #3 tablets required | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Allan Slomovic, MD, Principal Investigator — Toronto Western Hospital, University of Toronto
Locations (1):
- Toronto Western Hospital, University of Toronto, Toronto, Ontario, Canada